CLINICAL TRIAL: NCT06763042
Title: Evaluation of the Usability and Utility of Mindfulness-based Life Management Social Robots for Children and Adolescents in the Long-term Treatment Process
Brief Title: Usability and Utility of Mindfulness-based Life Management Social Robots for Children and Adolescents in the Long-term Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-03-057-006
Record Dates: First submitted 2023-08-30; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Cancer; Psychology, Child
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Groups that use the Mindfulness-based Life Management Social Robots (Experimental): Intervention period: 15-20 minutes or more per day for 14 days (at least 10 times in 2 weeks)
  Content: Life management content for mindfulness play and disease understanding
  Method of provision: Robot interaction using chatbot and remote conversation (mindfulness-based living management content and remote content will be provided for a total of 15 to 20 minutes)
  Interventions: Device: Mindfulness-based Life Management Social Robots

INTERVENTIONS:
Device: Mindfulness-based Life Management Social Robots — Mindfulness-based life management contents for pediatric patients operated by Social Robots

SUMMARY:
The purpose of this study is to apply social robot-based mindfulness-based life management content to pediatric and adolescent patients in the long-term disease treatment process and to assess usability and effectiveness of the social robot-based mindfulness-based life management content.

[Question 1] Effectiveness: Was the content on social robots effective in psychological adaptation of pediatric and adolescent patients?

[Question 2] Usability: Is there any difficulty in interacting through social robots applied in the hospital environment?

The participants conduct a preliminary survey and use robot content at least 10 times for the two weeks. Afterwards, follow-up surveys and in-depth interviews will be conducted.

DETAILED DESCRIPTION:
The purpose of this study is to apply social robot-based mindfulness-based life management content to pediatric and adolescent patients in the long-term disease treatment process and to assess usability and effectiveness of the social robot-based mindfulness-based life management content.

[Intervention]

* Intervention period: 15-20 minutes or more per day for 14 days (at least 10 times in 2 weeks)
* Content: Life management content for mindfulness play and disease understanding
* Method of provision: Robot interaction using chatbot and remote conversation (mindfulness-based living management content and remote content will be provided for a total of 15 to 20 minutes)

[Question 1] Effectiveness: Was the content on social robots effective in psychological adaptation of pediatric and adolescent patients?

(Measure) Pre-post comparison of survey result values

* Child Emotional and Behavioral Disorder Assessment Scale (Korea-Child Behavior Checklist: K-CBCL) ② Child and Youth Mindfulness Scale (Korean Child and Adolescent Mindfulness Measure: K-CAMM) ③ Child and Youth Optimism Scale (The Children's Life Orientation Test: C-LOT)

[Question 2] Usability: Is there any difficulty in interacting through social robots applied in the hospital environment?

(Measure) User Experience Questionnaire(UEQ), In-depth Interview

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6 to 12 years old who is being treated after the diagnosis of a severe or chronic disease
* Pediatric patients who need hospital treatment, including inpatient or outpatient treatment, for more than 3 months
* Pediatric patients with a level of communication that can be understood and agreed to in this study

Exclusion Criteria:

* Those who disagree with this study
* Pediatric patients who are judged to be difficult to interact with robots due to communication difficulties
* Pediatric patients who has been diagnosed with or is being treated for mental illness with psychotic characteristics

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluation Scale of Child Emotional and Behavioral Disorders | 14 days
  Measure and compare the score of Korea-Child Behavior Checklist (K-CBCL) before and after intervention. Change in psychological adaptation scores among pediatric and adolescent patients as measured by a validated psychological adaptation questionnaire. The questionnaire includes subscales for emotional regulation, coping mechanisms, and social engagement. Results will be reported as mean changes in scores from baseline to 14 days.
Measurement of Mindfulness Scale for Children and Adolescents | 14 days
  Measure and compare the score of Korean Child and Adolescent Mindfulness Measure (K-CAMM) before and after intervention. Change in psychological adaptation scores among pediatric and adolescent patients as measured by a validated psychological adaptation questionnaire. The questionnaire includes subscales for emotional regulation, coping mechanisms, and social engagement. Results will be reported as mean changes in scores from baseline to 14 days.
Measurement of optimism in children and adolescents | 14 days
  Measure and compare the score of The Children's Life Orientation Test (CLOT) before and after intervention. Change in psychological adaptation scores among pediatric and adolescent patients as measured by a validated psychological adaptation questionnaire. The questionnaire includes subscales for emotional regulation, coping mechanisms, and social engagement. Results will be reported as mean changes in scores from baseline to 14 days.

SECONDARY OUTCOMES:
Measurement of Measurement User Experience Questionnaire Short Version (UEQs) | 14 days
  Measurement of Measurement User Experience Questionnaire Short Version (UEQs) after intervention. Number of reported difficulties in interacting with the social robot, as assessed by a semi-structured usability survey. The survey includes items on ease of interaction, clarity of instructions, and overall user satisfaction. Responses will be quantified on a Likert scale (1 = very difficult, 5 = very easy).
In-depth interview | 14 days
  Interviews with study subjects based on the overall contents of the study

CONTACTS AND LOCATIONS:
Overall Officials: Meong Hi Son, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Centre, Seoul, Seoul, South Korea